CLINICAL TRIAL: NCT04618211
Title: A Phase II, Double-blind, Placebo-controlled, Randomized, Cross-over, Dose-ranging Study of Oral PHA-022121 for Acute Treatment of Angioedema Attacks in Patients With Hereditary Angioedema Due to C1-inhibitor Deficiency Type I and II
Brief Title: Dose-ranging Study of Oral PHA-022121 for Acute Treatment of Angioedema Attacks in Patients With Hereditary Angioedema
Acronym: RAPIDe-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharvaris Netherlands B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHA022121-C201; 2020-003445-11 (EudraCT Number)
Record Dates: First submitted 2020-10-26; First posted 2020-11-05 (Actual); Results first posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Angioedema; Hereditary Angioedema Type I; Hereditary Angioedema Type II; Hereditary Angioedema Types I and II; Hereditary Angioedema Attack; Hereditary Angioedema With C1 Esterase Inhibitor Deficiency; Hereditary Angioedema - Type 1; Hereditary Angioedema - Type 2; C1 Esterase Inhibitor Deficiency; C1 Inhibitor Deficiency
Keywords: HAE; HAE Type I; HAE Type II; Oral Treatment; Bradykinin B2 Receptor Antagonists; PHVS416; PHA121; PHA-022121; Deucrictibant
MeSH Terms: conditions — Angioedemas, Hereditary; Hereditary Angioedema Types I and II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose/placebo (Other): Single low dose of deucrictibant or placebo
  Interventions: Drug: Deucrictibant; Drug: Placebo
- Medium dose/placebo (Other): Single medium dose of deucrictibant or placebo
  Interventions: Drug: Deucrictibant; Drug: Placebo
- High dose/placebo (Other): Single high dose of deucrictibant or placebo
  Interventions: Drug: Deucrictibant; Drug: Placebo

INTERVENTIONS:
Drug: Deucrictibant — deucrictibant soft capsules for oral use
  Other Names: PHA-022121; PHA121; PHVS416
Drug: Placebo — Matching placebo capsules for oral use

SUMMARY:
This study evaluates the efficacy of orally administered deucrictibant for the acute treatment of attacks in patients with hereditary angioedema (HAE). Eligible subjects are randomized to one of three single doses of deucrictibant and placebo. The study will compare symptom relief (skin pain, skin swelling, abdominal pain) during HAE attacks and safety of each dose of deucrictibant with placebo.

DETAILED DESCRIPTION:
In Part I of the study, patients in non-attack state receive the assigned active single dose of deucrictibant at the study center to assess pharmacokinetics (the way the body absorbs, distributes, and gets rid of the drug) and safety. In Part II of the study, patients self-administer blinded study drug at home to treat three HAE attacks with deucrictibant or placebo (cross-over).

ELIGIBILITY:
Key Inclusion Criteria:

1. Signed and dated informed consent form
2. Diagnosis of HAE type I or II
3. Documented history of HAE attacks: at least three in the last 4 months, or at least two in the last 2 months prior to screening
4. Reliable access and experience to use standard of care acute attack medications

Key Exclusion Criteria:

1. Pregnancy or breast-feeding
2. Clinically significant abnormal electrocardiogram
3. Any other systemic disease or significant disease or disorder that would interfere with the patient's safety or ability to participate in the study
4. Use of C1-esterase inhibitor, oral kallikrein inhibitors, attenuated androgens, anti-fibrinolytics, or monoclonal HAE therapy within a defined period prior to enrollment
5. Positive serology for HIV or active infection with hepatitis B virus or hepatitis C virus
6. Abnormal hepatic function
7. Abnormal renal function
8. History of alcohol or drug abuse within defined period, or current evidence of substance dependence or abuse
9. History of documented severe hypersensitivity to any medicinal product
10. Participation in any other investigational drug study within defined period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Maurer, Prof MD, Principal Investigator — Charite University, Berlin, Germany
Locations (36):
- United States (8):
  - Study site, Birmingham, Alabama
  - Study site, Paradise Valley, Arizona
  - Study site, San Diego, California
  - Study site, Santa Monica, California
  - Study site, Walnut Creek, California
  - Study site, Chevy Chase, Maryland
  - Study site, St Louis, Missouri
  - Study site, Hershey, Pennsylvania
- Study site, Sofia, Bulgaria
- Canada (5):
  - Study site, Edmonton, Alberta
  - Study site, Ottawa, Ontario
  - Study site, Toronto, Ontario
  - Study site, Montreal, Quebec
  - Study site, Québec, Quebec
- Czechia (2):
  - Study site, Brno
  - Study site, Hradec Králové
- France (3):
  - Study site, Grenoble
  - Study site, Montpellier
  - Study site, Paris
- Germany (5):
  - Study site, Berlin
  - Study site, Dresden
  - Study site, Frankfurt
  - Study site, Mainz
  - Study site, Ulm
- Study site, Budapest, Hungary
- Israel (3):
  - Study site, Ashkelon
  - Study site, Haifa
  - Study site, Tel Aviv
- Italy (2):
  - Study site, Monserrato
  - Study site, Naples
- Study site, Amsterdam, Netherlands
- Study site, Krakow, Poland
- Spain (2):
  - Study site, Barcelona
  - Study site, Madrid
- United Kingdom (2):
  - Study site, Brighton
  - Study site, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 89 patients were screened, of which 74 patients were enrolled and randomized to the 3 PHA-022121 cohorts as follows: 25 participants to the 30 mg cohort, 25 participants to the 20 mg cohort, and 24 participants to the 10 mg cohort. From Part I to Part II, participants remained at their randomly assigned dose level. The majority of screen failures were due to inclusion criterion not met.
Pre-assignment Details: In Part I, participants in a quiescent state received a single dose of PHA-022121 at the assigned dose (10, 20, or 30 mg) to assess PK and safety. In Part II, participants received 2 single doses of PHA-022121 (10, 20, or 30 mg) and one single dose of placebo to assess efficacy and safety. Each participant administered their randomly assigned dose (either 10, 20, or 30 mg) for each of the 3 qualifying HAE attacks according to 1 of the 3 randomly assigned treatment sequences (crossover design).
Groups:
- PHA-022121 Low Dose - 10 mg: Part I: Single low dose of PHA-022121 (10 mg), non-attack state.
  Part II: 2 single low doses of PHA-022121 (10 mg) and one single dose of placebo in a 3-way crossover design, administered in the following sequence:
  1. Low dose / Low dose / Placebo
  2. Low dose / Placebo / Low dose
  3. Placebo / Low dose / Low dose
  Participants in Part I assigned to the Low Dose cohort remain in the Low Dose cohort in Part II.
- PHA-022121 Medium Dose - 20 mg: Part I: Single medium dose of PHA-022121 (20 mg), non-attack state.
  Part II: 2 single medium doses of PHA-022121 (20 mg) and one single dose of placebo in a 3-way crossover design:
  1. Medium dose / Medium dose / Placebo
  2. Medium dose / Placebo / Medium dose
  3. Placebo / Medium dose / Medium dose
  Participants in Part I assigned to the Medium Dose cohort remain in the Medium Dose cohort in Part II.
- PHA-022121 High Dose - 30 mg: Part I: Single high dose of PHA-022121 (30 mg), non-attack state.
  Part II: 2 single high doses of PHA-022121 (30 mg) and one single dose of placebo in a 3-way crossover design:
  1. High dose / High dose / Placebo
  2. High dose / Placebo / High dose
  3. Placebo / High dose / High dose
  Participants in Part I assigned to the High Dose cohort remain in the High Dose cohort in Part II.
Period: Part I (Non-Attack, Safety)
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg
Started | 24 | 25 | 25
Completed | 24 | 24 | 25
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Period: Part II (Self-administration, Efficacy)
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg
Started | 24 | 24 | 25
Attack 1 - PHA-022121 | 16 | 13 | 17
Attack 1 - Placebo | 6 | 6 | 6
Attack 2 - PHA-022121 | 12 | 8 | 12
Attack 2 - Placebo | 7 | 8 | 7
Attack 3 - PHA-022121 | 11 | 10 | 10
Attack 3 - Placebo | 7 | 3 | 6
Completed | 16 | 12 | 12
Not Completed | 8 | 12 | 13
Not completed — Withdrawal by Subject | 2 | 3 | 5
Not completed — Participants Met Primary Analysis Criteria | 6 | 9 | 8

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The FAS was defined as all participants enrolled and randomized in the study. Participants were analyzed based on the intention-to-treat principle, i.e., according to their randomized treatment assignment regardless of actual treatment taken.
Groups:
- PHA-022121 Low Dose - 10 mg: Part I: Single low dose of PHA-022121 (10 mg), non-attack state.
- PHA-022121 Medium Dose - 20 mg: Part I: Single medium dose of PHA-022121 (20 mg), non-attack state.
- PHA-022121 High Dose - 30 mg: Part I: Single high dose of PHA-022121 (30 mg), non-attack state.
- Total: Total of all reporting groups
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Total
Number analyzed (Participants) | 24 | 25 | 25 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (14.15) | 45.7 (13.89) | 41.4 (15.38) | 43.3 (14.41)
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 22 | 24 | 23 | 69
  From 65-84 years | 2 | 1 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 15 | 49
  Male | 7 | 8 | 10 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 22 | 24 | 25 | 71
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0
  Other | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 0 | 5
  Not Hispanic or Latino | 18 | 22 | 24 | 64
  Not Reported | 3 | 1 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change of the 3-symptom Composite Visual Analogue Scale (VAS-3) Score From Pre-treatment to 4 Hours Post-treatment
Description: The primary endpoint of the study was the change of the VAS-3 (3-symptom composite visual analogue scale) score from pre-treatment to 4 hours post-treatment. The VAS-3 was calculated as the mean of the VAS scores of the 3 major HAE symptoms: skin swelling, skin pain, and abdominal pain. The VAS scores of the 3 major HAE symptoms (skin swelling, skin pain, and abdominal pain) could range between 0 (No swelling/No pain) and 100 (Extreme swelling/Excruciating pain)
Time Frame: Assessed from pre-treatment to 4 hours post-treatment
Population: Part I efficacy data not collected, consistent with and pre-specified in the study protocol. Includes all participants with evaluable data who completed the relevant assessment time point.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- PHA-022121 Low Dose - 10 mg: Part II: 2 single low doses of PHA-022121 (10 mg) and one single dose of placebo in a 3-way crossover design:
  1. Low dose / Low dose / Placebo
  2. Low dose / Placebo / Low dose
  3. Placebo / Low dose / Low dose
  Part II efficacy data utilized for the analysis.
- PHA-022121 Medium Dose - 20 mg: Part II: 2 single medium doses of PHA-022121 (20 mg) and one single dose of placebo in a 3-way crossover design:
  1. Medium dose / Medium dose / Placebo
  2. Medium dose / Placebo / Medium dose
  3. Placebo / Medium dose / Medium dose
  Part II efficacy data utilized for the analysis.
- PHA-022121 High Dose - 30 mg: Part II: 2 single high doses of PHA-022121 (30 mg) and one single dose of placebo in a 3-way crossover design:
  1. High dose / High dose / Placebo
  2. High dose / Placebo / High dose
  3. Placebo / High dose / High dose
  Part II efficacy data utilized for the analysis.
- Placebo: Part II: 2 single high doses of PHA-022121 (10, 20, or 30 mg) and one single dose of placebo in a 3-way crossover design:
  1. PHA-022121 dose / PHA-022121 dose / Placebo
  2. PHA-022121 dose / Placebo / PHA-022121 dose
  3. Placebo / PHA-022121 dose / PHA-022121 dose
  Part II efficacy data utilized for the analysis.
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Score on a scale | -14.83 (1.833) | -13.10 (2.111) | -14.37 (1.975) | 1.92 (1.596)
Statistical Analysis 1: Comparison: PHA-022121 Low Dose - 10 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed model repeated measures — Nominal p-value; Least squares mean difference = -16.75, 95% CI 2-sided [-21.52 to -11.97], Standard Error of Mean 2.423
Statistical Analysis 2: Comparison: PHA-022121 Medium Dose - 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed model repeated measures; Least squares mean difference = -15.02, 95% CI 2-sided [-20.22 to -9.81], Standard Error of Mean 2.64
Statistical Analysis 3: Comparison: PHA-022121 High Dose - 30 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed model repeated measures; Least squares mean difference = -16.28, 95% CI 2-sided [-21.27 to -11.29], Standard Error of Mean 2.531

2. Secondary Outcome: Time to Onset of Symptom Relief by ≥30% Reduction in Visual Analogue Scale (VAS-3) Composite Score From the Pre-treatment Score
Description: VAS-3 scores range between 0 and 100.
Time Frame: Assessed from pre-treatment to 48-hours post-treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Groups:
- PHA-022121 Low Dose -10 mg: Part II: 2 single low doses of PHA-022121 (10 mg) and one single dose of placebo in a 3-way crossover design:
  1. Low dose / Low dose / Placebo
  2. Low dose / Placebo / Low dose
  3. Placebo / Low dose / Low dose
  Part II efficacy data utilized for the analysis.
Arm/Group | PHA-022121 Low Dose -10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Hours | 2.1 [1.5 to 2.9] | 2.7 [1.9 to 3.5] | 2.5 [1.9 to 3.8] | 8.0 [7.6 to 48.0]
Statistical Analysis 1: Comparison: PHA-022121 Low Dose -10 mg; Test type: Superiority; p < 0.0001, Marginal Cox Proportional Hazards Model — Nominal p-value; Hazard Ratio (HR) = 3.81, 95% CI 2-sided [2.01 to 7.2]
Statistical Analysis 2: Comparison: PHA-022121 Medium Dose - 20 mg; Test type: Superiority; p = 0.0021, Marginal Cox Proportional Hazards Model; Hazard Ratio (HR) = 3.08, 95% CI 2-sided [1.5 to 6.3]
Statistical Analysis 3: Comparison: PHA-022121 High Dose - 30 mg; Test type: Superiority; p < 0.0001, Marginal Cox Proportional Hazards Model; Hazard Ratio (HR) = 3.61, 95% CI 2-sided [2.1 to 6.19]

3. Secondary Outcome: Time to Onset of Almost Complete or Complete Symptom Relief by Visual Analogue Scale (VAS-3)
Description: VAS scores range between 0 and 100. Almost complete symptom relief is defined as all 3 individual VAS scores of the VAS-3 having a value < 10. Complete symptom relief is defined as all 3 individual VAS scores are of the VAS-3 having a value of 0.
Time Frame: Assessed from pre-treatment to 48 hours post-treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Hours | 5.8 [3.6 to 7.5] | 20.0 [4.5 to 20.0] | 20.0 [6.0 to 20.1] | 42.0 [22.0 to 48.0]
Statistical Analysis 1: Comparison: PHA-022121 Low Dose - 10 mg vs Placebo; Test type: Superiority; p < 0.0001, Cox Proportional Hazards Model — Nominal p-value; Hazard Ratio (HR) = 5.09, 95% CI 2-sided [2.81 to 9.22]
Statistical Analysis 2: Comparison: PHA-022121 Medium Dose - 20 mg vs Placebo; Test type: Superiority; p = 0.0127, Marginal Cox Proportional Hazards Model; Hazard Ratio (HR) = 2.25, 95% CI 2-sided [1.19 to 4.27]
Statistical Analysis 3: Comparison: PHA-022121 High Dose - 30 mg vs Placebo; Test type: Superiority; p = 0.0001, Marginal Cox Proportional Hazards Model; Hazard Ratio (HR) = 2.65, 95% CI 2-sided [1.61 to 4.38]

4. Secondary Outcome: Time to a ≥50% Reduction in VAS-3 Composite Score From the Pre-treatment Score
Description: Time to a ≥50% reduction in VAS-3 composite score from the pre-treatment score.
Time Frame: Assessed from pre-treatment to 48 hours post-treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Hours | 3.3 [2.4 to 3.9] | 4.0 [2.9 to 6.0] | 4.0 [3.3 to 5.8] | 22.8 [20.0 to 24.1]
Statistical Analysis 1: Comparison: PHA-022121 Low Dose - 10 mg vs Placebo; Test type: Superiority; p < 0.0001, Marginal Cox Proportional Hazards Model — Nominal p-value; Hazard Ratio (HR) = 4.55, 95% CI 2-sided [2.41 to 8.59]
Statistical Analysis 2: Comparison: PHA-022121 Medium Dose - 20 mg vs Placebo; Test type: Superiority; p = 0.0003, Marginal Cox Proportional Hazards Model; Hazard Ratio (HR) = 3.65, 95% CI 2-sided [1.8 to 7.38]
Statistical Analysis 3: Comparison: PHA-022121 High Dose - 30 mg vs Placebo; Test type: Superiority; p < 0.0001, Marginal Cox Proportional Hazards Model; Hazard Ratio (HR) = 3.87, 95% CI 2-sided [2.26 to 6.63]

5. Secondary Outcome: Change in the Mean Symptom Complex Severity (MSCS) Score From Pre-treatment to 4 Hours Post-treatment
Description: MSCS scores range between 0 and 3. A higher score means a worse outcome.
Time Frame: Pre-treatment and 4 hours post-treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Score on a scale | -1.08 [-1.33 to -0.83] | -0.91 [-1.19 to -0.62] | -0.68 [-0.95 to -0.40] | -0.29 [-0.51 to -0.08]
Statistical Analysis 1: Comparison: PHA-022121 Low Dose - 10 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed model repeated measures — Nominal p-value; Least squares mean difference = -0.79, 95% CI 2-sided [-1.11 to -0.46], Standard Error of Mean 0.164
Statistical Analysis 2: Comparison: PHA-022121 Medium Dose - 20 mg vs Placebo; Test type: Superiority; p = 0.0008, Mixed model repeated measures; Least squares mean difference = -0.61, 95% CI 2-sided [-0.97 to -0.26], Standard Error of Mean 0.178
Statistical Analysis 3: Comparison: PHA-022121 High Dose - 30 mg vs Placebo; Test type: Superiority; p = 0.0291, Mixed model repeated measures; Least squares mean difference = -0.39, 95% CI 2-sided [-0.73 to -0.04], Standard Error of Mean 0.174

6. Secondary Outcome: Treatment Outcome Score (TOS) at 4 Hours Post-treatment
Description: TOS range between -100 and 100. A positive score indicates improvement, a score of 0 indicates no change, and a negative score indicates worsening compared to pre-treatment.
Time Frame: 4 hours post-treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Score on a scale | 60.52 [41.74 to 79.29] | 59.08 [37.58 to 80.57] | 67.44 [47.15 to 87.74] | -3.62 [-19.68 to 12.45]
Statistical Analysis 1: Comparison: PHA-022121 Low Dose - 10 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed model repeated measures — Nominal p-value; Least squares mean difference = 64.13, 95% CI 2-sided [40.35 to 87.91], Standard Error of Mean 12.016
Statistical Analysis 2: Comparison: PHA-022121 Medium Dose - 20 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed model repeated measures; Least squares mean difference = 62.69, 95% CI 2-sided [36.71 to 88.67], Standard Error of Mean 13.128
Statistical Analysis 3: Comparison: PHA-022121 High Dose - 30 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed model repeated measures; Least squares mean difference = 71.06, 95% CI 2-sided [46.09 to 96.03], Standard Error of Mean 12.613

7. Secondary Outcome: Time to Onset of Primary Symptom Relief Assessed by a 30% Reduction in the VAS for the Primary Symptom
Description: Time to onset of primary symptom relief assessed by a 30% reduction in the VAS for the primary symptom within 48 hours post-treatment
Time Frame: Within 48 hours post-treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Hours | 2.0 [1.4 to 2.4] | 3.0 [1.9 to 4.1] | 2.9 [1.9 to 3.9] | 23.3 [6.1 to NA] — Insufficient number of participants with events.

8. Secondary Outcome: Proportion of Study Drug Treated Attacks Requiring HAE Rescue Medication Within 12 Hours.
Description: Proportion of blinded study drug treated attacks requiring HAE rescue medication within 12 hours post-treatment.
Time Frame: Assessed at 12 hours post study drug treatment
Population: as for outcome 1
Measure: Number; unit: Attacks requiring HAE rescue medication
Units Other Than Participants: Number of Treated Attacks
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Number analyzed (Number of Treated Attacks) | 37 | 28 | 31 | 51
Attacks requiring HAE rescue medication | 7 | 3 | 2 | 31

9. Secondary Outcome: Time to First HAE Rescue Medication Use for Study Drug-treated Attacks Within 48 Hours Post-treatment
Description: The proportion of treated attacks with first use of HAE rescue medication within 48 hours post-treatment with PHA-022121.
Time Frame: Assessed at 48 hours post study drug treatment
Population: Part I efficacy data not collected, consistent with and pre-specified in the study protocol. Includes all participants with evaluable data who completed the relevant assessment time point. Medians are as follows: Low Dose 10 mg - NA (
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Hours | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | NA [NA to NA] — Insufficient number of participants with events. | 6.0 [4.4 to 13.1]

10. Secondary Outcome: Time to Change in the VAS Score for Skin Pain Score - 30% Reduction
Description: Time to change in the VAS score for Skin Pain Score - 30% reduction within 48-hours post-treatment. VAS-3 scores range between 0 and 100. A larger reduction means a better outcome.
Time Frame: Within 48 hours post treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 17 | 10 | 17 | 34
Hours | 2.9 [1.9 to 5.7] | 3.4 [1.9 to 6.0] | 2.7 [1.9 to 3.9] | 22.8 [8.7 to NA] — Insufficient number of participants with events.

11. Secondary Outcome: Change in Mean Symptom Complex Severity Score From Pre-treatment to 24 Hours Post-treatment
Description: Change in the Mean Symptom Complex Severity (MSCS) score from pre-treatment to 24 hours post-treatment. A lower MSCS score indicates a better outcome.
Time Frame: 24 hours post-treatment
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Score on a scale | -1.65 (0.117) | -1.50 (0.123) | -1.68 (0.122) | -1.20 (0.163)

12. Secondary Outcome: TOS at 24 Hours Post-treatment
Description: Treatment outcome score at 24 hours post-treatment. A higher score indicates improvement.
Time Frame: Assessed within 24 hours post treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Score on a scale | 94.44 (21.183) | 93.60 (21.190) | 94.44 (16.013) | 76.92 (38.813)

13. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication Scores at 48 Hours Post-treatment - Effectiveness Domain Score
Description: MMRM analysis of Treatment Satisfaction Questionnaire for Medication (TSQM) at 48 hours post-treatment. The 11-item TSQM (version II) evaluated participant treatment satisfaction with the medication for the following scales: effectiveness, side effects, convenience, and overall satisfaction Scale scores were transformed into scores ranging from 0 to 100 and could be used to calculate a total composite score, a higher score indicating greater satisfaction.
Time Frame: 48 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Score on a scale | 79.17 (23.179) | 70.45 (30.290) | 72.92 (23.085) | 65.38 (23.532)

14. Secondary Outcome: Time to Onset of Primary Symptom Relief by 50% Reduction in VAS Score
Description: Time to Onset of Primary Symptom Relief by 50% Reduction in VAS Score within 48 hours post-treatment. VAS-3 scores range between 0 and 100. A larger reduction means a better outcome.
Time Frame: Within 48 hours post-treatment
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Hours | 2.9 [2.4 to 3.9] | 4.5 [2.9 to 8.5] | 4.0 [2.5 to 5.8] | 22.8 [5.8 to 24.1]

15. Secondary Outcome: Proportion of Study Drug Treated Attacks Requiring HAE Rescue Medication Within 24 Hours.
Description: Qualifying attacks treated with study drug may use approved rescue medication if no symptom relief within 4 hours has been experienced.
Time Frame: Assessed at 24 hours post-study drug treatment
Population: as for outcome 1
Measure: Number; unit: Attacks requiring HAE rescue medication
Units Other Than Participants: Number of Treated Attacks
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Number analyzed (Number of Treated Attacks) | 37 | 28 | 31 | 51
Attacks requiring HAE rescue medication
  Number of treated attacks | 37 | 28 | 31 | 51
  Number of treated attacks requiring HAE rescue medication | 9 | 3 | 4 | 37

16. Secondary Outcome: Proportion of Study Drug Treated Attacks Requiring HAE Rescue Medication Within 48 Hours
Description: as for outcome 15
Time Frame: Assessed at 48 hours post-study drug treatment
Population: as for outcome 1
Measure: Number; unit: Attacks requiring HAE rescue medication
Units Other Than Participants: Number of Treated Attacks
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Number analyzed (Number of Treated Attacks) | 37 | 28 | 31 | 51
Attacks requiring HAE rescue medication
  Number of treated attacks | 37 | 28 | 31 | 51
  Number of treated attacks requiring HAE rescue medication | 9 | 4 | 5 | 37

17. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication Scores at 48 Hours Post-treatment - Convenience Domain Score
Description: as for outcome 13
Time Frame: 48 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Score on a scale | 80.56 (16.569) | 83.08 (23.096) | 77.55 (20.229) | 76.07 (27.441)

18. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication Scores at 48 Hours Post-treatment - Satisfaction Domain Score
Description: as for outcome 13
Time Frame: 48 hours post-treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 21 | 16 | 20 | 51
Score on a scale | 82.50 (18.907) | 80.68 (29.702) | 76.74 (22.113) | 64.10 (24.623)

19. Secondary Outcome: Time to Change in the VAS Score for Skin Swelling Score - 30% Reduction
Description: Time to change in the VAS score for Skin Swelling Score - 30% reduction within 48 hours post-treatment. VAS-3 scores range between 0 and 100. A larger reduction means a better outcome.
Time Frame: Within 48 hours post-treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 17 | 12 | 18 | 40
Hours | 2.5 [1.4 to 5.8] | 3.5 [2.2 to 20.0] | 3.8 [1.9 to 4.8] | 23.3 [3.9 to NA] — Insufficient number of participants with events.

20. Secondary Outcome: Time to Change in the VAS Score for Abdominal Pain Score - 30% Reduction
Description: Time to change in the VAS score for Abdominal Pain Score - 30% reduction within 48 hours post-treatment. VAS-3 scores range between 0 and 100. A larger reduction means a better outcome.
Time Frame: Within 48 hours post-treatment
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | PHA-022121 Low Dose - 10 mg | PHA-022121 Medium Dose - 20 mg | PHA-022121 High Dose - 30 mg | Placebo
Number analyzed (Participants) | 12 | 8 | 9 | 20
Hours | 1.9 [1.1 to 2.1] | 1.4 [0.9 to 2.5] | 2.9 [1.9 to 7.5] | 20.0 [2.9 to NA] — Insufficient number of participants with events.

ADVERSE EVENTS:
Time Frame: All AEs (including SAEs) recorded from the time of signing informed consent until the end-of-study visit. Timeframe for reporting adverse events: 5 days post-treatment.
Description: Adverse events are reported separately for Part I (non-attack) and Part II within the table below, as in Part I, study participants administered a single dose of study drug to assess PK and safety, and in Part II, study participants administered study drug to treat up to 3 qualified HAE attacks.
  For Part II, total participants at risk and total number of attacks at risk are reported separately. Part II total participants at risk reflect randomized treatment assignments and pooled attacks.
Groups:
- Part I PHA-022121 Low Dose - 10 mg: Part I: Single low dose of PHA-022121 (10 mg), non-attack state.
- Part I PHA-022121 Medium Dose - 20 mg: Part I: Single medium dose of PHA-022121 (20 mg), non-attack state.
- Part I PHA-022121 High Dose - 30 mg: Part I: Single high dose of PHA-022121 (30 mg), non-attack state.
- Part II PHA-022121 Low Dose - 10 mg Study Drug Treated Attacks: Part II: 2 single low doses of PHA-022121 (10 mg) and one single dose of placebo in a 3-way crossover design:
  1. Low dose / Low dose / Placebo
  2. Low dose / Placebo / Low dose
  3. Placebo / Low dose / Low dose
  Number at risk reflects number of study drug treated attacks.
- Part II PHA-022121 Medium Dose - 20 mg Study Drug Treated Attacks: Part II: 2 single medium doses of PHA-022121 (20 mg) and one single dose of placebo in a 3-way crossover design:
  1. Medium dose / Medium dose / Placebo
  2. Medium dose / Placebo / Medium dose
  3. Placebo / Medium dose / Medium dose
  Number at risk reflects number of study drug treated attacks.
- Part II PHA-022121 High Dose - 30 mg Study Drug Treated Attacks: Part II: 2 single high doses of PHA-022121 (30 mg) and one single dose of placebo in a 3-way crossover design:
  1. High dose / High dose / Placebo
  2. High dose / Placebo / High dose
  3. Placebo / High dose / High dose
  Number at risk reflects number of study drug treated attacks.
- Part II PHA-022121 Low Dose - 10 mg Participants: Part II: 2 single low doses of PHA-022121 (10 mg) and one single dose of placebo in a 3-way crossover design:
  1. Low dose / Low dose / Placebo
  2. Low dose / Placebo / Low dose
  3. Placebo / Low dose / Low dose
  Number at risk reflects number of participants at risk.
- Part II PHA-022121 Medium Dose - 20 mg Participants: Part II: 2 single medium doses of PHA-022121 (20 mg) and one single dose of placebo in a 3-way crossover design:
  1. Medium dose / Medium dose / Placebo
  2. Medium dose / Placebo / Medium dose
  3. Placebo / Medium dose / Medium dose
  Number at risk reflects number of participants at risk.
- Part II PHA-022121 High Dose - 30 mg Participants: Part II: 2 single high doses of PHA-022121 (30 mg) and one single dose of placebo in a 3-way crossover design:
  1. High dose / High dose / Placebo
  2. High dose / Placebo / High dose
  3. Placebo / High dose / High dose
  Number at risk reflects number of participants at risk.
- Part II Placebo: Part II: 2 single high doses of PHA-022121 (10, 20, or 30 mg) and one single dose of placebo in a 3-way crossover design:
  1. PHA-022121 dose / PHA-022121 dose / Placebo
  2. PHA-022121 dose / Placebo / PHA-022121 dose
  3. Placebo / PHA-022121 dose / PHA-022121 dose
Arm/Group | Part I PHA-022121 Low Dose - 10 mg | Part I PHA-022121 Medium Dose - 20 mg | Part I PHA-022121 High Dose - 30 mg | Part II PHA-022121 Low Dose - 10 mg Study Drug Treated Attacks | Part II PHA-022121 Medium Dose - 20 mg Study Drug Treated Attacks | Part II PHA-022121 High Dose - 30 mg Study Drug Treated Attacks | Part II PHA-022121 Low Dose - 10 mg Participants | Part II PHA-022121 Medium Dose - 20 mg Participants | Part II PHA-022121 High Dose - 30 mg Participants | Part II Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24 | 0/25 | 0/38 | 0/29 | 0/36 | 0/21 | 0/16 | 0/22 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24 | 0/25 | 0/38 | 0/29 | 0/36 | 0/21 | 0/16 | 0/22 | 0/53
Other Adverse Events (participants affected / at risk) | 2/23 | 2/24 | 4/25 | 3/38 | 1/29 | 2/36 | 3/21 | 1/16 | 2/22 | 4/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I PHA-022121 Low Dose - 10 mg (N=23) | Part I PHA-022121 Medium Dose - 20 mg (N=24) | Part I PHA-022121 High Dose - 30 mg (N=25) | Part II PHA-022121 Low Dose - 10 mg Study Drug Treated Attacks (N=38) | Part II PHA-022121 Medium Dose - 20 mg Study Drug Treated Attacks (N=29) | Part II PHA-022121 High Dose - 30 mg Study Drug Treated Attacks (N=36) | Part II PHA-022121 Low Dose - 10 mg Participants (N=21) | Part II PHA-022121 Medium Dose - 20 mg Participants (N=16) | Part II PHA-022121 High Dose - 30 mg Participants (N=22) | Part II Placebo (N=53)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mean cell hemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mean cell volume decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Primary analysis is presented. For the endpoints "Time to Onset of Symptom Relief by 30% Reduction in Visual Analogue Scale (VAS-3)," "Time to almost or complete symptom relief by VAS," & "Time to 50% reduction in VAS-3," the within participant correlation was not accounted for in the Kaplan-Meier estimation of median time and corresponding 95% confidence interval.

Participant flow is reported according to randomized treatment cohort, efficacy & safety results are according to treatment group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT04618211/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT04618211/SAP_001.pdf